CLINICAL TRIAL: NCT04647695
Title: An Open-label Randomized Controlled Trial on Interferon β-1b and Remdesivir Combination Versus Remdesivir as Treatment for COVID-19 Infection
Brief Title: IFN-beta 1b and Remdesivir for COVID19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 20-535
Record Dates: First submitted 2020-11-27; First posted 2020-12-01 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: COVID-19; IFN-beta 1b; remdesivir; hospitalised
MeSH Terms: conditions — COVID-19 | interventions — Interferon beta-1b; remdesivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IFN-beta 1b and remdesivir (Experimental): a 5-day course of subcutaneous injection of interferon β-1b 2mL (16 million IU) consecutively and IV remdesivir 200mg loading on day 1 followed by remdesivir 100mg daily on day 2 to day 5
  Interventions: Drug: Interferon beta-1b
- Remdesivir (Active Comparator): a 5-day course of IV remdesivir 200mg loading on day 1 followed by remdesivir 100mg daily on day 2 to day 5
  Interventions: Drug: Remdesivir

INTERVENTIONS:
Drug: Interferon beta-1b — a 5-day course of subcutaneous injection of interferon β-1b 2mL (16 million IU) consecutively and IV remdesivir 200mg loading on day 1 followed by remdesivir 100mg daily on day 2 to day 5
  Other Names: Remdesivir
  Arms: IFN-beta 1b and remdesivir
Drug: Remdesivir — a 5-day course of IV remdesivir 200mg loading on day 1 followed by remdesivir 100mg daily on day 2 to day 5
  Arms: Remdesivir

SUMMARY:
A 5-day combination of interferon β-1b and remdesivir will expedite the recovery, suppress the viral load and shorten hospitalisation in patients with SARS-CoV-2 infection compare to the control arm

DETAILED DESCRIPTION:
Introduction The novel coronavirus (SARS-CoV-2), is a single-stranded RNA coronavirus. The virus was first isolated from patients presented with pneumonia in Wuhan in December 2019. It is believed that the virus first emerged from patients working in the Wuhan Seafood Market which also sold contaminated wild animals, consumed as a local delicacy. Sequences of the Wuhan betacoronavirus show similarities to betacoronaviruses found in bats, sharing a common ancestor with the 2003 SARS coronavirus (SARS-CoV) and the bat coronavirus HKU, a virus found in fruit bats. Similar to SARS-CoV, it is a member of Beta-CoV lineage B. Five genomes of the novel coronavirus have been initially isolated and reported including BetaCoV/Wuhan/IVDC-HB-01/2019, BetaCoV/Wuhan/IVDC-HB-04/2020, BetaCoV/Wuhan/IVDC-HB-05/2019, BetaCoV/Wuhan/WIV04/2019, and BetaCoV/Wuhan/IPBCAMS-WH-01/2019 from the China CDC.

The SARS-CoV-2 has since spread from China to the rest of the world. As of 20 November 2020, more than 50 million people been confirmed to have infected by SARS-CoV-2, resulting in more than 1,000,000 deaths. Remdesivir has been shown to clinically effective in severe Covid-19 patients but virological data is lacking. FDA has approved the use of remdesivir for the treatment of severe Covid-19 infection. Apart from remdesivir, no specific antiviral treatment for the SARS-CoV-2 is currently available, but existing medication could be repurposed.

Genetic sequencing demonstrated similarity of the SARS-CoV-2 to the SARS-CoV and MERS CoV. We expect patients infected with the SARS-CoV-2 will also present similarly with initial upper respiratory tract symptoms including fever, cough, sputum, myalgia and shortness or breath. More severe cases might complicate with pneumonia and required ventilatory or ECMO support. According to our previous studies in 2003 on patients hospitalized for severe SARS-CoV, the viral load peaked between day 7 from symptoms onset and coincided with clinical deterioration of pneumonia and respiratory failure, with majority of the patients required intensive care support. Higher viral load isolated from different human system also correlated with worsened SARS manifestation and complications.

Previously, the investigators have demonstrated that interferon-beta1b, commonly used in the treatment of multiple sclerosis and lopinavir/ ritonavir, also demonstrated to improve the outcome of MERS-CoV infection in a non-human primate model of common marmoset. A more recent open-label, randomized controlled trial by our team has proven that interferon beta-1b, in combination with lopinavir/ ritonavir and ribavirin reduced the SARS-CoV-2 viral load in the respiratory tract and resulted in faster alleviation of clinical symptoms when compared to lopinavir/ ritonavir alone or with ribavirin, suggesting that interferon beta-1b was likely to be the backbone of this triple therapy.

Therefore, the investigators propose to conduct an open-label randomized controlled trial on interferon beta-1b and remdesivir combination versus remdesivir as treatment for patients hospitalized for COVID-19 infection

Patients will be randomly assigned to one of the two groups: Group A: a 5-day course of subcutaneous injection of interferon β-1b 2mL (16 million IU) consecutively and IV remdesivir 200mg loading on day 1 followed by remdesivir 100mg daily on day 2 to day 5, or Group B: a 5-day course of IV remdesivir 200mg loading on day 1 followed by remdesivir 100mg daily on day 2 to day 5 (1:1).

ELIGIBILITY:
Inclusion Criteria:

1. Recruited subjects include all adult patients ≥18 years hospitalized for virologic confirmed SARS-CoV-2 infection.
2. Fulfilling one of the following criteria associated with high risk of clinical deterioration: age 65 years or above, radiological evidence of pneumonia, oxygen desaturation <94% on room air, comorbidity including hypertension, diabetes, cardiovascular diseases, chronic obstructive lung disease, chronic liver diseases, chronic kidney diseases, malignancy, haematological diseases, rheumatological diseases, immunocompromised hosts and obesity (BMI > 30)
3. All subjects give written informed consent. For patients who are critically ill, requiring ICU, ventilation or confused, informed consent will be obtained from spouse, next-of-kin or legal guardians.
4. Subjects must be available to complete the study and comply with study procedures. Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

1. Inability to comprehend and to follow all required study procedures.
2. Allergy or severe reactions to the study drugs
3. Patients taking medication that will potentially interact with l interferon beta-1b and remdesivir
4. Patients with known history of severe depression
5. Estimated glomerular filtration rate <30 mL/min
6. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to recruitment in this study or expect to receive an experimental agent during this study.
7. To participate in an unrelated trial during the current clinical trial. Nevertheless, the patients have the right to withdraw from the current clinical trial to join another clinical trial.
8. Have a history of alcohol or drug abuse in the last 5 years.
9. Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 30 days
  Time to complete alleviation of symptoms as defined by NEWS of 0 maintained for 24 hours

SECONDARY OUTCOMES:
Hospitalisation | 30 days
  Length of hospitalization
NPS viral load | 7 days
  Time to negative nasopharyngeal swab (NPS) SARS-CoV-2 RT-PCR
TS viral load | 7 days
  Time to negative throat saliva (TS) SARS-CoV-2 RT-PCR
Inflammatory markers | 7 days
  Cytokine/ chemokine changes
Adverse events | 5 days
  Adverse events during treatment
Mortality | 30 days
  30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Anonymous IPD will be shared upon request to the HKU IRB and approved by the panel
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon study publication for 12 months
Access Criteria: Approval by the IRB panel

REFERENCES:
- [Background] Blanco-Melo D, Nilsson-Payant BE, Liu WC, Uhl S, Hoagland D, Moller R, Jordan TX, Oishi K, Panis M, Sachs D, Wang TT, Schwartz RE, Lim JK, Albrecht RA, tenOever BR. Imbalanced Host Response to SARS-CoV-2 Drives Development of COVID-19. Cell. 2020 May 28;181(5):1036-1045.e9. doi: 10.1016/j.cell.2020.04.026. Epub 2020 May 15. PMID 32416070
- [Background] Chu H, Chan JF, Wang Y, Yuen TT, Chai Y, Hou Y, Shuai H, Yang D, Hu B, Huang X, Zhang X, Cai JP, Zhou J, Yuan S, Kok KH, To KK, Chan IH, Zhang AJ, Sit KY, Au WK, Yuen KY. Comparative Replication and Immune Activation Profiles of SARS-CoV-2 and SARS-CoV in Human Lungs: An Ex Vivo Study With Implications for the Pathogenesis of COVID-19. Clin Infect Dis. 2020 Sep 12;71(6):1400-1409. doi: 10.1093/cid/ciaa410. PMID 32270184
- [Background] Yuan S, Chan CC, Chik KK, Tsang JO, Liang R, Cao J, Tang K, Cai JP, Ye ZW, Yin F, To KK, Chu H, Jin DY, Hung IF, Yuen KY, Chan JF. Broad-Spectrum Host-Based Antivirals Targeting the Interferon and Lipogenesis Pathways as Potential Treatment Options for the Pandemic Coronavirus Disease 2019 (COVID-19). Viruses. 2020 Jun 10;12(6):628. doi: 10.3390/v12060628. PMID 32532085
- [Background] Chan JF, Yao Y, Yeung ML, Deng W, Bao L, Jia L, Li F, Xiao C, Gao H, Yu P, Cai JP, Chu H, Zhou J, Chen H, Qin C, Yuen KY. Treatment With Lopinavir/Ritonavir or Interferon-beta1b Improves Outcome of MERS-CoV Infection in a Nonhuman Primate Model of Common Marmoset. J Infect Dis. 2015 Dec 15;212(12):1904-13. doi: 10.1093/infdis/jiv392. Epub 2015 Jul 21. PMID 26198719
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Result] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440
- [Result] Hung IF, Lung KC, Tso EY, Liu R, Chung TW, Chu MY, Ng YY, Lo J, Chan J, Tam AR, Shum HP, Chan V, Wu AK, Sin KM, Leung WS, Law WL, Lung DC, Sin S, Yeung P, Yip CC, Zhang RR, Fung AY, Yan EY, Leung KH, Ip JD, Chu AW, Chan WM, Ng AC, Lee R, Fung K, Yeung A, Wu TC, Chan JW, Yan WW, Chan WM, Chan JF, Lie AK, Tsang OT, Cheng VC, Que TL, Lau CS, Chan KH, To KK, Yuen KY. Triple combination of interferon beta-1b, lopinavir-ritonavir, and ribavirin in the treatment of patients admitted to hospital with COVID-19: an open-label, randomised, phase 2 trial. Lancet. 2020 May 30;395(10238):1695-1704. doi: 10.1016/S0140-6736(20)31042-4. Epub 2020 May 10. PMID 32401715
- [Derived] Tam AR, Zhang RR, Lung KC, Liu R, Leung KY, Liu D, Fan Y, Lu L, Lam AH, Chung TW, Yip CC, Lo J, Wu AK, Lee R, Sin S, Ng PY, Chan WM, Shum HP, Yan WW, Chan JF, Cheng VC, Lau CS, To KK, Chan KH, Yuen KY, Hung IF. Early Treatment of High-Risk Hospitalized Coronavirus Disease 2019 (COVID-19) Patients With a Combination of Interferon Beta-1b and Remdesivir: A Phase 2 Open-label Randomized Controlled Trial. Clin Infect Dis. 2023 Feb 8;76(3):e216-e226. doi: 10.1093/cid/ciac523. PMID 35762834